CLINICAL TRIAL: NCT03547336
Title: A Randomized, Controlled, Open-label, Parallel Study in End Stage Renal Disease (ESRD) Patients on Hemodialysis Comparing the Theranova Dialyzer to Hemodiafiltration
Brief Title: Study in End Stage Renal Disease (ESRD) Patients on Hemodialysis Comparing the Theranova Dialyzer to Hemodiafiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7408001
Record Dates: First submitted 2018-05-16; First posted 2018-06-06 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theranova 400 Dialyzer (Experimental): In-center hemodialysis (in HD mode), 3 times a week for 12 week duration. The patient will undergo regular HD treatment on the first treatment of the first week of study, after which, the patient will switch to the randomized dialyzer, from the second treatment to the end of study treatment. Blood sampling will be obtained at the hospital by trained personnel according to local routines.
  Interventions: Device: Theranova 400 Dialyzer
- FX800 (Active Comparator): In-center hemodialysis (in HDF mode), 3 times a week for 12 week duration. The patient will undergo regular HD treatment on the first treatment of the first week of study, after which, the patient will switch to the randomized dialyzer, from the second treatment to the end of study treatment. Blood sampling will be obtained at the hospital by trained personnel according to local routines.
  Interventions: Device: FX800 Dialyzer

INTERVENTIONS:
Device: Theranova 400 Dialyzer — Dialysis performed in HD mode. Treatment duration for each individual subject will vary based on clinical requirements determined by the Investigator, based on the subject's need, residual renal function, access function, tolerance to HD/HDF and other relevant factors. The participating subjects' HD/HDF prescriptions should be kept stable throughout the study.
  Arms: Theranova 400 Dialyzer
Device: FX800 Dialyzer — Dialysis performed in HDF mode. Treatment duration for each individual subject will vary based on clinical requirements determined by the Investigator, based on the subject's need, residual renal function, access function, tolerance to HD/HDF and other relevant factors. The participating subjects' HD/HDF prescriptions should be kept stable throughout the study.
  Arms: FX800

SUMMARY:
In China, the estimated prevalence of patients with ESRD receiving PD or maintenance HD increased from 51.7 per million population (pmp) at the end of 2007 to 79.1 pmp at the end of 2008. Theranova 400 is designed to deliver the performance of hemodiafiltration (HDF) using standard hemodialysis (HD) equipment and treatment mode, including HD machines, disposables, blood and dialysate flows, length of treatment and frequency of treatment. Theranova 400 utilizes a Medium Cut-Off (MCO) membrane with extended permeability for middle solutes to closely modulate the removal function of the kidney without the complexity of HDF. The primary objective of the study is to demonstrate non-inferiority of the Theranova Dialyzer in hemodialysis (HD) mode compared to hemodiafiltration (HDF), using FX 800 in HDF mode. Comparison of the study arms over time will be used to support the safety of Theranova 400 by demonstrating stable serum albumin levels, as well as support the dialyzer's efficacy to significantly remove serum middle molecules.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients who are able to give IC after an explanation of the proposed study.
* Patients who have Kt/Vurea > 1.2 for the last 2 measurements, with the most recent Kt/Vurea measurement taken within 4 weeks before or during study screening.
* Patients with a dialysis prescription (dialyzer, time, dialysis fluid flow rate (QD), blood flow rate (QB)) stable over 6 recent treatments. The dialysis treatment time should be 3.5 to 4.5 hours per session with minimum QB of at least 250 mL/min and QD of 500 mL/min.
* Patients who are on stable anticoagulation prescription and dose.
* Patients with ESRD receiving chronic HD treatment with a history of thrice weekly HD, and at least 1 HDF session within 1 month prior to study.
* Patients who have been stable on in-center HD for >3 months prior to study enrollment
* Patients who have an adequate arteriovenous (AV) fistula or graft, or dual-lumen tunneled catheter capable of providing a blood flow rate of at least 250 mL/min.
* Patients with a minimum total convective volume (including ultrafiltration (UF)) of 16 L post-dilution for the most recent HDF treatment.
* Patients who receive in-center treatment hemodialysis at a site that routinely implements high flux dialysis and HDF.

Exclusion Criteria:

* Patients who have acute renal failure with the chance for recovery.
* Patients who are pre-scheduled for a living donor kidney transplant within the next six months, who plan a change to PD within the next six months, or who require single-needle dialysis therapy.
* Pregnant and lactating women.
* Patients with positive serology tests for Hepatitis B surface antigen, Hepatitis C total antibody), HIV and Syphilis.
* Patients with known hemodynamic instability, anemia (Hgb < 90 g/L), and/or patients with Hgb >130g/L for coagulation risk.
* Patients who are severely malnourished or with significant disease that interferes with liver synthetic function, e.g. with serum albumin <35 g/L.
* Patients with active or ongoing infection as per investigator's judgement.
* Patients with history of solid tumors requiring anti-cancer therapy in the past or next 6 months, or life expectancy less than 1 year, or patients or with history of hematology neoplasm.
* Patients diagnosed with a NYHA Class IV congestive heart failure, or acute coronary syndrome and/or who have suffered a myocardial infarction within three months prior to the start of the study.
* Patients with a history of severe mental disorders.
* Patients who are currently participating in, or have previously participated in other interventional clinical trials during the past 4 weeks.
* Patients who have had an allergic response to polyarylethersulfone (PAES) or polysulfone (PS) membrane or have history of poor tolerance to dialyzers with synthetic membranes
* Patients with advanced liver, heart or pulmonary disease as judged by the Investigator.
* Patients with any comorbidity possibly conflicting with the study purpose or procedures as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-01-04 (Actual)

PRIMARY OUTCOMES:
Reduction ratio of lambda free light chains (λ FLC) | Up to 1 week
  At the first mid-week treatment day
Reduction ratio of β2 microglobulin | Up to 1 week
  At the first mid-week treatment day
Pre-dialysis serum albumin | Study Completion (Week 12)

SECONDARY OUTCOMES:
Kt/V urea | Week 1, Week 5, Week 9, Week 13
  Mid-Week Treatment Day
Urea reduction ratio (URR) | Week 1, Week 5, Week 9, Week 13
  Mid-Week Treatment Day
Pre-dialysis serum levels of λ FLC | Week 1, Week 5, Week 9, Week 13
  Mid-Week Treatment Day
Pre-dialysis serum levels of β2 microglobulin | Week 1, Week 5, Week 9, Week 13
  Mid-Week Treatment Day
Reduction ratio of α1 microglobulin (α1M) | Up to 1 week
  At the first mid-week treatment day
Reduction ratio of Chitinase-3-like protein (YKL-40) | Up to 1 week
  At the first mid-week treatment day
Reduction ratio of complement factor D (CFD) | Up to 1 week
  At the first mid-week treatment day
Reduction ratio of myoglobin | Up to 1 week
  At the first mid-week treatment day
Reduction ratio of kappa free light chains (κ FLC) | Up to 1 week
  At the first mid-week treatment day

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Investigational Site, Hefei, Anhui
  - Investigational Site, Guangzhou, Guangdong
  - Investigational Site, Zhengzhou, Henan
  - Investigational Site, Wuhan, Hubei
  - Investigational Site, Shanghai, Shanghai Municipality
  - Investigational Site, Chengdu, Sichuan
  - Investigational Site, Hangzhou, Zhejiang
  - Investigational Site, Beijing